CLINICAL TRIAL: NCT05490056
Title: Adequacy of Antenatal Care and Its Determinants in Assiut District
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marwa Fazzaa Hassan Farag, Physician at Egyptian Ministry of Health and Population, Assiut University
Other Study IDs: Adequacy of ANC in Assiut
Record Dates: First submitted 2022-08-01; First posted 2022-08-05 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-03

CONDITIONS: Maternal Care Patterns
Keywords: antenatal care

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — the study will not apply on intervention

SUMMARY:
Cross sectional study on women who gave birth and attend immunization session for their children in Assiut District to assess the adequacy of ANC, its determinants and knowledge and attitude of antenatal care among the studied women

DETAILED DESCRIPTION:
The World health organization (WHO) estimated that worldwide in 2021, about 211 women died per 100,000 live birth from pregnancy related causes and increasing to 415 on average in the poorest countries (1)Globally in 2020, nearly 2.4 million babies died during the first 28 days of life (2). High coverage of quality Antenatal Care (ANC) can play a crucial role to decrease maternal and child mortality rates and achieve national and global targets related to maternal and child health. ANC received from skilled provider increases maternal and newborn survival and reduces the risk of pregnancy complications and adverse pregnancy outcomes(3) .

New WHO guidelines on antenatal care for a positive pregnancy experience include:

1. A minimum of eight contacts are recommended.
2. Counselling about healthy eating and keeping physically active during pregnancy.
3. Daily oral iron and folic acid supplementation
4. Tetanus toxoid vaccination is recommended.
5. One ultrasound scan before 24 weeks' gestation.
6. Health-care providers should ask all pregnant women about their use of alcohol and other substances(4).

The 2016 WHO prenatal care guidelines for a healthy pregnancy experience reflect a change from the centered ANC model with a prescribed minimum of 4 ANC visits (ANC4+) to a more expanded model that emphasizes contact number, timing, and services(5). At the global and national levels, most currently available data indicate that women receive at least 4 antenatal care visits. There is very limited data on the adequacy of ANC based and their correlates on updated WHO recommendations for antenatal care(5, (6),(7)). The current study is conducted in accordance with the research plan of Public Health and Community Medicine Department- Faculty of Medicine, Assiut University.

ELIGIBILITY:
Inclusion Criteria :

women of reproductive age who gave birth

-

Exclusion Criteria:

Pregnant and menopaused women

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — women of reproductive age who gave birth
Study Population: This study will be carried on women gave birth and come to immunize their children aged 2 months. The selection of index mother will be done during children vaccination sessions as the high vaccination coverage in Egypt give higher opportunity for non- biased selection of the studied population.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-02-01 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Adequacy of ANC | 2 years
  ): Adequacy of ANC among women who gave birth and attend immunization sessions for their children in Assiut District and its determinants based on receiving all the following 11 ANC items at least once:
  * adequate number of ANC visits (at least 8 ANC visits)
  * early ANC use (1st ANC booking during 1st trimester)
  * Provision of ANC by a skilled provider (doctor or trained nurse).
  * Measurement of blood pressure
  * A blood sample was taken
  * urine sample was taken
  * Receiving tetanus toxoid
  * Weight measurement
  * Ultrasound was performed
  * Being informed about danger signs of pregnancy
  * And receiving health education about nutrition and prescription oral iron and folic acid supplements.

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Attia, Professor, Principal Investigator — Assiut Universiyy

REFERENCES:
- [Result] Osterman MJK, Martin JA. Timing and Adequacy of Prenatal Care in the United States, 2016. Natl Vital Stat Rep. 2018 May;67(3):1-14. PMID 29874159
- [Result] Pugliese-Garcia M, Radovich E, Hassanein N, Campbell OMR, Khalil K, Benova L. Temporal and regional variations in use, equity and quality of antenatal care in Egypt: a repeat cross-sectional analysis using Demographic and Health Surveys. BMC Pregnancy Childbirth. 2019 Jul 26;19(1):268. doi: 10.1186/s12884-019-2409-1. PMID 31349804
- [Result] El Aty MA, Meky FA, Morsy M, El Sayed MK. Overall adequacy of antenatal care in Oman: secondary analysis of national reproductive health survey data, 2008. East Mediterr Health J. 2015 Feb 2;20(12):781-8. PMID 25664516
- See also: New guidelines on antenatal care for a positive pregnancy experience — http://www.who.int/news/item/07-11-2016-new-guidelines-on-antenatal-care-for-a-positive-pregnancy-experience
- See also: https://www.who.int/news/item/05-10-2021-new-global-targets-to-prevent-maternal-deaths — https://www.who.int/news/item/05-10-2021-new-global-targets-to-prevent-maternal-deaths